CLINICAL TRIAL: NCT01518894
Title: A Randomized, Double-Blind, Placebo Controlled, Sponsor Open, Phase 1b Study To Examine The Safety, Tolerability And Pharmacokinetics Of PF-04958242 In Psychiatrically Stable Subjects With Schizophrenia
Brief Title: A Study To Examine The Safety, Tolerability And Pharmacokinetics Of PF-04958242 In Psychiatrically Stable Subjects With Schizophrenia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: B1701004
Record Dates: First submitted 2012-01-23; First posted 2012-01-26 (Estimated); Last update posted 2019-11-21 (Actual); Status verified 2019-11

CONDITIONS: Schizophrenia
Keywords: PF-04958242; multiple dose; Safety; schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — PF-04958242

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- PF-04958242 (Experimental)
  Interventions: Drug: PF-04958242
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PF-04958242 — PF-04958242 0.10 mg oral solution Q24 hours for 14 days
  Arms: PF-04958242
Drug: PF-04958242 — PF-04958242 0.20 mg oral solution Q24 hours for 14 days
  Arms: PF-04958242
Drug: PF-04958242 — PF-04958242 oral solution Q24 hours for 14 days (dose to be determined)
  Arms: PF-04958242
Drug: Placebo — Placebo oral solution Q24 hours for 14 days
  Arms: Placebo

SUMMARY:
To evaluate the safety and tolerability of multiple, ascending doses of PF-04958242 administered orally to psychiatrically stable subjects with schizophrenia receiving antipsychotic and adjunctive medication.

DETAILED DESCRIPTION:
This study was previously posted by Pfizer, Inc. Sponsorship of the trial was transferred to Biogen.

ELIGIBILITY:
Inclusion Criteria:

* Psychiatrically stable subjects with schizophrenia
* Evidence of stable schizophrenia symptomatology ≥ 3 months
* Score on MCCB Letter-number span + Spatial span subtest < 40.

Exclusion Criteria:

* History of seizures or of a condition with risk of seizures
* History of abnormal EEG.
* Pregnant or nursing females, and women of child bearing potential

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2011-11; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Composite of Pharmacokinetics measured at 0.25, 0.5, 0.75, 1, 2, 3, 4, 8, 12, 24 hours after dosing on Day 1 | Day 1 - Day 2
Composite of Pharmacokinetics measured pre-dose and 1 hour post-dose on Day 4 | Day 4
Composite of Pharmacokinetics measured pre-dose and 1 hour post-dose on Day 7 | Day 7
Composite of Pharmacokinetics measured at 0.25, 0.5, 0.75, 1, 2, 3, 4, 8, 12, 24, 48, 72, 120 hours after dosing on Day 14 | Day 14 - Day 17
Composite of urine Pharmacokinetics measured for 24 hours post-dose on Day 14 | Day 14 - Day 15

SECONDARY OUTCOMES:
Cogntion - CogState | Day 0, 1, 6, 13
Cognition - Matrics Consensus Cognition Battery | Day 0, 1, 6, 13
Drug Effect Questionnaire liking scale | Day, 1, 14
Cognitive training | Days 0 - 13
Columbia Suicide Severity Rating Scale | Day 0, 1, 7, 14, 17, 23

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (1):
- Pfizer Investigational Site, Long Beach, California, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1701004&StudyName=A%20Study%20To%20Examine%20The%20Safety%2C%20Tolerability%20And%20Pharmacokinetics%20Of%20%20PF-04958242%20In%20Psychiatrically%20Stable%20Subjects%20With%20Schizophrenia